CLINICAL TRIAL: NCT02853071
Title: Efficacy and Safety of Estracyt® in Metastatic Breast Cancer Hormonal Estrogen Receptor (HER 2) Negative, Hormone Receptor (HR) Positive.
Brief Title: Efficacy and Safety of Estracyt® in Metastatic Breast Cancer
Acronym: BEST
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: withdrawal industrial
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P/2015/269
Record Dates: First submitted 2016-07-29; First posted 2016-08-02 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Estramustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Estramustine (Experimental): 560 mg per day
  Interventions: Drug: Estramustine
- Standard practice center (Active Comparator): Standard treatment center choice.
  Excepted: anthracyclines, taxanes, capecitabine and eribulin
  Interventions: Drug: standard practice

INTERVENTIONS:
Drug: Estramustine
  Other Names: estracyt, estramustine phosphate
  Arms: Estramustine
Drug: standard practice — standard practice
  Arms: Standard practice center

SUMMARY:
This study evaluates efficacy, safety and quality of life in patients affected by metastatic breast cancer RH+/ HER2- and treated by estramustine phosphate.

DETAILED DESCRIPTION:
For patients affected by metastatic breast cancer RH+/HER2-, the conventional treatment is hormonotherapy. But, when patients don't react no recommendations exist.

Estramustine phosphate is currently prescribed for prostate cancer. The estramustine phosphate is an active anti-tumoral agent by oral route, associating a nitrogenous mustard with the estradiol, it settles on membrane receptor and the cytotoxic component acts essentially by dismantling microtubules inhibiting the mitosis.

Estramustine could be a therapeutic option when currently therapy are exhausted for patients reactive to hormonotherapy previous lines or chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic breast cancer HER2-/RH+
* Progression after hormonotherapy
* Treated by taxanes, anthracyclines, capecitabine and eribulin
* Treated by everolimus
* ECOG ≤ 2
* Hematological Function: neutrophiles ≥ 1,5 x 109 / L, hemoglobin ≥ 9 g / dL, plaques ≥ 100 x 109 / L
* Hepatic function: albumin ≥ 2,5 g / dl, bilirubin serum ≤ 2 x N (superior border of the standard) (unless disease of Gilbert), transaminases ≥ 3 x N
* Renal Function: serum creatinine ≤ 1,5 mg / dL or clearance of the creatinine ≥ 40 mL / min
* Estimated Life expectancy ≥ 3 months

Exclusion Criteria:

* Hypersensitivity known about one of the constituents of the estramustine phosphates
* Preliminary Treatment by estramustine phosphates
* Brain Metastases
* Patients not being under effective contraception
* Minor, pregnant or lactating Patients
* Patients not previously treated by everolimus
* Transaminases > 3xN
* Other concomitant anticancer treatment less than 1 month before the inclusion
* Digestive function: malabsorption
* History of other cancer in the previous 5 years (other than squamous-cell epithelioma or totally resected in situ carcinoma)
* Active Thrombo-phlebitis
* Risk thromboembolic known,
* Unchecked cardiovascular Pathology
* Grave hepatic Affection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of the alive patients without progress of the disease | 3 months

SECONDARY OUTCOMES:
quality of life | 18 months
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 items (EORTC QLQ-C30)
progression-free survival | 18 months
overall survival | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Régional Universitaire, Besançon, France

IPD SHARING:
Plan to Share IPD: Yes
The Committee shall meet twice a year